CLINICAL TRIAL: NCT02656043
Title: A Phase 1 and 2 Randomized, Double-Blind, Vehicle-Controlled, Parallel-Group Study to Evaluate the Safety, Tolerability, Efficacy, and Exposure of up to 12 Weeks of XPF-005 Treatment in Healthy Volunteers and Subjects With Acne Vulgaris
Brief Title: A Safety, Tolerability, Efficacy and Exposure Study of XEN801 Topical Gel
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Xenon Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: XPF-005-101
Record Dates: First submitted 2016-01-12; First posted 2016-01-14 (Estimated); Last update posted 2019-01-22 (Actual); Status verified 2019-01

CONDITIONS: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- XPF-005 (Active Comparator): Active treatment: XPF-005 Gel
  Interventions: Drug: XPF-005
- Vehicle gel (Placebo Comparator): Placebo: XPF-005 Vehicle Gel
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: XPF-005 — Comparison of active treatment XPF-005 topical gel against Placebo (XPF-005 Vehicle Gel) applied to face for acne vulgaris.
  Arms: XPF-005
Drug: Placebo
  Arms: Vehicle gel

SUMMARY:
Phase 1/2 study enrolling up to 60 healthy volunteers in Phase 1 followed by approximately 150 subjects with acne vulgaris in Phase 2.

DETAILED DESCRIPTION:
Phase 1/2 study enrolling up to 60 healthy volunteers followed by approximately 150 subjects with acne vulgaris. Data from Phase 1 stage will be reviewed before progressing to Phase 2.

Phase 1 is an open label study to determine safety, tolerability of XPF-005 topical gel and exposure of XEN801 (active ingredient). Up to 5 cohorts of 12 healthy volunteers will each receive different dose volumes of XPF-005 gel or Placebo gel on their face and back for 14 or 21 days. Safety assessments are completed and PK samples are collected at study visits.

Phase 2 is a randomized, double-blind, vehicle-controlled, parallel-group study to determine safety, tolerability, efficacy of XPF-005 topical gel and exposure of XEN801 (active ingredient). Approximately 150 subjects with acne vulgaris will apply XPF-005 or matching placebo gel on their face for 12 weeks. Safety and efficacy assessments are completed and PK samples are collected at study visits.

Safety assessments include local skin tolerability assessments, vital signs, physical examination, 12-lead ECG, safety laboratory blood and urine and adverse event reporting.

Efficacy assessments include acne lesion counts and Investigator's Global Assessment (IGA).

ELIGIBILITY:
Key Inclusion Criteria:

1. Aged between 18 and 50, inclusive
2. Male or female, agree to comply with contraceptive requirements
3. Signed Informed Consent Form
4. Clinical diagnosis of facial acne vulgaris defined as:

   * 25 to 75 inflammatory lesions,
   * 20 to 120 non-inflammatory lesions, and
   * an IGA score of ≥3
5. Agree to refrain from using any topical acne treatments on the face or any oral acne treatments. Topical acne treatment that do not have significant or measurable systemic absorption are permitted for treatment of the back, shoulders, and chest only

Key Exclusion Criteria:

1. Known sensitivity to any topical or dermal product, including alcohol
2. Female who is breast feeding, pregnant, or planning to become pregnant
3. Any skin condition of the face other than acne vulgaris
4. Two or more active nodular lesions
5. Excessive facial hair that would interfere with the evaluation of safety or with the diagnosis or assessment of acne vulgaris
6. Use of tanning beds/booths, or excessive sun exposure
7. Use of over-the-counter topical medications for treatment of acne vulgaris on the face within 14 days of baseline
8. Use of systemic corticosteroids, antibiotics, anti-acne drugs, anti-inflammatory drugs (NSAIDs are permitted) or prescription topical retinoid use on the face within 28 days prior the baseline
9. Initiation of hormonal therapy or dose change to hormonal therapy within 12 weeks prior to baseline.
10. Use of androgen receptor blockers (eg, spironolactone, flutamide) within 12 weeks prior to baseline
11. Use of oral retinoid (eg, isotretinoin, alitretinoin) within 12 months prior to baseline and vitamin A supplements >10,000 units/day within 6 months prior to baseline
12. Facial procedures (eg, microdermabrasion, chemical or laser peel) within 8 weeks prior to baseline
13. Photodynamic therapy within 12 weeks prior to baseline
14. Any other reason that would make the subject, in the opinion of the Investigator or Sponsor, unsuitable for the study

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 213 (Actual)
Dates: Start 2015-09-17 (Actual); Primary Completion 2017-02-16 (Actual); Study Completion 2017-03-17 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in acne lesion count | Week 12

SECONDARY OUTCOMES:
Change from Baseline in acne lesion count | Week 4 and 8
Change from Baseline in Investigator Global Assessment (IGA) | Week 4, 8 and 12

CONTACTS AND LOCATIONS:
Overall Officials: Xenon Pharmaceuticals Inc., Study Director — Xenon Pharmaceuticals Inc.
Locations (20):
- Canada (20):
  - Kirk Barber Research, Calgary, Alberta
  - Institute for Skin Advancement, Calgary, Alberta
  - Stratica Medical Inc., Edmonton, Alberta
  - Dr. Chih-ho Hong Medical Inc., Surrey, British Columbia
  - Carruthers & Humphrey Clinical Research, Vancouver, British Columbia
  - Pacific Dermaesthetics, Vancouver, British Columbia
  - Toole Dermatology Research, Winnipeg, Manitoba
  - Clinique Médicale Nepisiguit, Bathurst, New Brunswick
  - SimcoDerm Medical and Surgical Dermatology Center, Barrie, Ontario
  - Lynderm Research Inc, Markham, Ontario
  - DermEdge Research, Mississauga, Ontario
  - Research by ICLS, Oakville, Ontario
  - York Dermatology Center, Richmond Hill, Ontario
  - Bayview North Dermatology Clinic, Toronto, Ontario
  - G. Daniel Schachter Medicine Professional Corporation, Toronto, Ontario
  - K. Papp Clinical Research Inc, Waterloo, Ontario
  - Windsor Clinical Research Inc., Windsor, Ontario
  - Innovaderm Research Inc., Montreal, Quebec
  - Dre Angélique Gagné-Henley M.D. Inc, Saint-Jérôme, Quebec
  - Siena Medical Research Corporation, Westmount, Quebec